CLINICAL TRIAL: NCT00320801
Title: A Randomized, Double-Blind, Multicenter Study Evaluating The Safety and Efficacy of BTDS in Subjects With Moderate to Severe Osteoarthritis Pain. Includes a 52-Week Extension Phase.
Brief Title: Buprenorphine Transdermal Patches (BTDS) in Subjects With Osteoarthritis Pain. Includes a 52-week Extension Phase.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to administrative reasons.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3014 and BUP3014S; NCT01137422 (obsolete NCT alias)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Chronic pain; osteoarthritis; transdermal
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BTDS 5 (Active Comparator): Buprenorphine transdermal patch 5 mcg/h, applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal patch
- BTDS 20 (Experimental): Buprenorphine transdermal patch 20 mcg/h, applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
  Other Names: Butrans™
  Arms: BTDS 5
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
  Other Names: Butrans™
  Arms: BTDS 20

SUMMARY:
The original objective of this study was to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (BTDS) 20 micrograms (mcg)/hour (h) in comparison to the buprenorphine transdermal system 5 mcg/h in subjects with moderate to severe osteoarthritis pain currently treated with oral opioids. The double-blind treatment intervention duration is 12 weeks during which time supplemental analgesic medication (acetaminophen or ibuprofen) will be provided to all subjects in addition to study drug.

This study was terminated early due to administrative reasons with only 20% of the planned sample size; therefore, the primary objective was changed to focus on the safety evaluation.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the hip, knee, or spine for 1 year or longer.
* taking between 30-80 milligrams (mg) of oral morphine sulfate or equivalent/day, at least 4 days a week.

Exclusion Criteria:

* taking more than 80 mg per day of oral morphine sulfate or equivalent within 30 days of enrollment.
* requiring frequent analgesic therapy for chronic conditions in addition to osteoarthritis.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah O'Keefe, BSN, Study Chair — Purdue Pharma L.P., Stamford, CT
Locations (66):
- United States (66):
  - Parkway Medical Center, Birmingham, Alabama
  - Edwards Lake Medical Center, Birmingham, Alabama
  - Rheumatogogy Associates of N. Alabama,, Huntsville, Alabama
  - Drug Research and Analysis Corp., Montgomery, Alabama
  - Meadowbrook Research, Scottsdale, Arizona
  - Research Solutions, LLC, Searcy, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Crest Clinical Research, Inc, Anaheim, California
  - NuLife Clinical Research, Inc., Anaheim, California
  - Orange County Clinical Research, Cypress, California
  - Private Practice, Laguna Hills, California
  - Andwell Research, Laguna Niguel, California
  - Valerius Medical Group & Research Center Inc., Long Beach, California
  - Anesthesiology and Pain Management, Los Gatos, California
  - Scripps Clinic Ranchro Bernardo, San Diego, California
  - Orrin M. Troum & Medical Associates, Santa Monica, California
  - Diablo Clinical Research, Walnut Creek, California
  - Private Practice, Arvada, Colorado
  - Mountainview Clinical Research, Denver, Colorado
  - Private Practice, Aventura, Florida
  - Medical Research Associates, Clearwater, Florida
  - LifeSpan Clinical Research, Miami, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Family Practice of St. Cloud PA Wilker/Powers Center for Clinical Studies, Saint Cloud, Florida
  - Wilker/Powers Center for Clinical Studies, Saint Cloud, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - University Neurology, Sarasota, Florida
  - Pinnacle Trials, Inc., Atlanta, Georgia
  - Clinical Investigative Services Med College of Georgia, Augusta, Georgia
  - America's Doctor (SMO), Gurnee, Illinois
  - Dolby Providers, Inc., New Orleans, Louisiana
  - Professional Clinical Research, Cadillac, Michigan
  - Private Practice, Oak Park, Michigan
  - Lake Michigan Clinical Research and Consulting, Inc., Saint Joseph, Michigan
  - Research Center of the Ozarks, , MO, Everton, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Cherry Hill Orthopedic Surgeons, Cherry Hill, New Jersey
  - Private Practice, Medford, New Jersey
  - Univeristy of Medicine and Dentistry of New Jersey, Stratford, New Jersey
  - Crescent Medical Assoc., Astoria, New York
  - Private Practice, Plainview, New York
  - State University of NY at Stonybrook, Stony Brook, New York
  - Charlotte Spine Center Pain and Orthopedic Neurology, Pain Research Institute of the Carolinas, Charlotte, North Carolina
  - Albermarle Family Practice, Elizabeth City, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Odyssey Research Services, Bismarck, North Dakota
  - Midwest Regional Research, Bellbrook, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Lyle, Austin Alexander PA, Tulsa, Oklahoma
  - Rouge Valley Clinical Research, Medford, Oregon
  - Southern Oregon Health & Wellness, Medford, Oregon
  - Keystone Clinical Solutions, Inc., Altoona, Pennsylvania
  - Sidney Hillman Medical Center, Philadelphia, Pennsylvania
  - Arcuri Clinical Research, Philadelphia, Pennsylvania
  - The Arthritis & Osteoporosis Center, Orangeburg, South Carolina
  - Alpha Clinical Research, Clarksville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Integrity Clinical Research, LLC (SMO), Milan, Tennessee
  - LifeTree Clinical Reseach, Salt Lake City, Utah
  - J. Lewis Research Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research Foothill Family Clinic South, Salt Lake City, Utah
  - Arthritis Clinic of No. Virginia, Arlington, Virginia
  - MedSource, Richmond, Virginia
  - Vantage Clinical Research Group, Lacey, Washington
  - Arthritis Northwest, Seattle, Washington
  - Clinical Trials Northwest, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 07-Jan-2004 (First subject first visit); 09-Mar-2005 (last subject last visit of extension [subjects went directly into the extension upon completion of the double-blind phase]) at 42 sites in the United States (US).
Pre-assignment Details: Adult subjects (≥ 40 years), with osteoarthritis (OA) of the hip, knee or spine for longer than 1 year, controlled on oral opioid therapy, who met the inclusion/exclusion criteria specified in the protocol. The open-label run-in period (N = 188) selected subjects who tolerated BTDS 20 mcg/h and showed stable pain control (N = 96 completed).
Groups:
- Run-in Period: (≤14 days). The run-in period was designed to select subjects who tolerated and responded to BTDS 20. Subjects were eligible to enter the double-blind phase if they tolerated BTDS 20 and achieved stable analgesia.
- Double-blind BTDS 5: Reference treatment: Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
- Double-blind BTDS 20: Test treatment: buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
- Extension Phase: Subjects received open-label buprenorphine transdermal patch 5, 10 or 20 mcg/h applied for 7-day wear for up to 52 weeks.
Period: Open-label Run-in Period
Arm/Group | Run-in Period | Double-blind BTDS 5 | Double-blind BTDS 20 | Extension Phase
Started | 188 | 0 | 0 | 0
Completed | 96 | 0 | 0 | 0
Not Completed | 92 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0 | 0
Not completed — Administrative | 10 | 0 | 0 | 0
Not completed — Lack of Efficacy | 44 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Did not qualify | 1 | 0 | 0 | 0
Period: Double-blind Phase
Arm/Group | Run-in Period | Double-blind BTDS 5 | Double-blind BTDS 20 | Extension Phase
Started | 0 | 47 | 49 | 0
Completed | 0 | 36 | 35 | 0
Not Completed | 0 | 11 | 14 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 8 | 0
Not completed — Administrative | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 9 | 1 | 0
Period: Extension Phase
Arm/Group | Run-in Period | Double-blind BTDS 5 | Double-blind BTDS 20 | Extension Phase
Started | 0 | 0 | 0 | 55
Completed | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 48
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 8
Not completed — Administrative | 0 | 0 | 0 | 29
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Total
Number analyzed (Participants) | 47 | 49 | 96
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.65) | 61.1 (11.72) | 59.6 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 13 | 21 | 34

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events (AEs) as a Measure of Safety.
Description: Safety assessments included monitoring and recording of all adverse events and serious adverse events (SAEs).
Time Frame: Throughout BTDS exposure (Includes run-in period, double-blind phase and extension phase)
Population: The safety population consists of all subjects who received at least 1 dose of study drug and had at least 1 safety assessment after the initial dose of BTDS in the study.
Measure: Number; unit: Participants
Groups:
- Run-in Period: The run-in period was designed to determine tolerability of BTDS 20. Subjects were eligible to enter the double-blind phase if they tolerated BTDS 20 and achieved stable analgesia.
- Overall BTDS Exposure: Overall core and extension phase combined (run-in period, double-blind phase, and extension phase)
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Run-in Period | Overall BTDS Exposure
Number analyzed (Participants) | 47 | 49 | 188 | 188
Participants
  Deaths | 0 | 0 | 0 | 0
  Serious adverse events | 1 | 1 | 2 | 6
  Other Adverse Events in ≥ 4.5% of subjects | 17 | 22 | 52 | 101

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) that occurred after the signing of the informed consent up to end of study and 7 days after discontinuation, or Serious AEs occurring up to 30 days following the last study visit were followed until the AE resolved or stabilized.
Description: AEs were learned of by spontaneous reports, subject interview, and daily diary.
Groups:
- Double-blind BTDS 5: Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
- Double-blind BTDS 20: Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
- Open-label Run-in Period: The run-in period (14 days) was designed to identify subjects whose pain was controlled with and who tolerated BTDS 20. Open-label BTDS 10 or 20 mcg/h applied for 7-day wear to qualify for randomization into the double-blind phase.
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Open-label Run-in Period | Overall BTDS Exposure
Serious Adverse Events (participants affected / at risk) | 1/47 | 1/49 | 2/188 | 6/188
Other Adverse Events (participants affected / at risk) | 17/47 | 22/49 | 52/188 | 101/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS 5 (N=47) | Double-blind BTDS 20 (N=49) | Open-label Run-in Period (N=188) | Overall BTDS Exposure (N=188)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Systematic and nonsystematic assessments.
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Chest pressure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Somnolent (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Worsening of reflex sympathetic dystrophy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments.
Grade 2 splenic laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Right occipital condyle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Comminuted pelvic fracture left (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Right tibia-fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Sphenoid fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Comminuted acetabulum left (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Right lower lobe contusion on chest (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Left post distal shaft fibular fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Left lower lobe contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Subarachnoid hemorrhage of fourth ventricle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Left hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments.
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS 5 (N=47) | Double-blind BTDS 20 (N=49) | Open-label Run-in Period (N=188) | Overall BTDS Exposure (N=188)
Nausea (Gastrointestinal disorders) | 4 | 3 | 30 | 38 — Systematic and nonsystematic assessments.
Vomiting NOS (Gastrointestinal disorders) | 1 | 2 | 16 | 21 — Systematic and nonsystematic assessments.
Constipation (Gastrointestinal disorders) | 1 | 5 | 4 | 9 — Systematic and nonsystematic assessments.
Edema peripheral (General disorders) | 4 | 4 | 5 | 18 — Systematic and nonsystematic assessments.
Application site pruritus (General disorders) | 3 | 5 | 9 | 17 — Systematic and nonsystematic assessments.
Application site erythema (General disorders) | 3 | 5 | 4 | 14 — Systematic and nonsystematic assessments.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 3 | 16 — Systematic and nonsystematic assessments.
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 4 — Systematic and nonsystematic assessments.
Headache (Nervous system disorders) | 4 | 2 | 16 | 24 — Systematic and nonsystematic assessments.
Dizziness (Nervous system disorders) | 2 | 1 | 15 | 20 — Systematic and nonsystematic assessments.
Anxiety (Psychiatric disorders) | 3 | 0 | 1 | 5 — Systematic and nonsystematic assessments.
Application site rash (General disorders) | 2 | 1 | 7 | 15 — Systematic and nonsystematic assessments.
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 11 — Systematic and nonsystematic assessments.
Somnolence (Nervous system disorders) | 2 | 2 | 6 | 10 — Systematic and nonsystematic assessments.
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 9 — Systematic and nonsystematic assessments.

LIMITATIONS AND CAVEATS:
Study terminated due to administrative reasons. The primary objective was changed to a safety study prior to unblinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days